CLINICAL TRIAL: NCT02014311
Title: Myocardial Perfusion 320 MDCT Guided Treatment Strategy for the Clinical Management of Patient With Recent Acute-onset Chest Pain. A Randomized Controlled Trial
Brief Title: CArdiac cT in the Treatment of Acute CHest Pain 2 - Myocardial CT Perfusion
Acronym: CATCH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Amager Hospital (Other); Bispebjerg Hospital (Other); Herlev Hospital (Other); Glostrup University Hospital, Copenhagen (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Klaus Fuglsang Kofoed, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-3-2013-065
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease
Keywords: Multidetector Computed Tomography; Myocardial Perfusion Imaging; Coronary Stenosis; Coronary Artery Disease; Angina Pectoris
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Angina Pectoris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTA+CTP guided treatment strategy (Experimental): Patients with adenosine stress induced regional myocardial hypoperfusion (CT perfusion imaging) in combination with a corresponding epicardial coronary vessel with >50% stenosis (Coronary CT angiography) will be referred for invasive investigation within 30 days after study inclusion - CTP-INTERVENTION
  Interventions: Procedure: CTA+CTP guided treatment strategy
- CTA guided treatment strategy (Active Comparator): Patients with at least one epicardial coronary artery stenosis >50% (Coronary CT angiography) will be referred for invasive investigation within 30 days after initial discharge from the hospital - CONTROL
  Interventions: Procedure: CTA guided treatment strategy

INTERVENTIONS:
Procedure: CTA+CTP guided treatment strategy — CTA+CTP guided treatment strategy
  Arms: CTA+CTP guided treatment strategy
Procedure: CTA guided treatment strategy — CTA guided treatment strategy
  Arms: CTA guided treatment strategy

SUMMARY:
The aim of this study is to assess whether the clinical management of patients with recent acute-onset chest pain without acute coronary syndrome may be optimized by a combined coronary CT angiography (CTA) + CT myocardial perfusion (CTP) guided, rapid diagnostic strategy as compared to CTA alone. CT diagnostic evaluation and potential referral for invasive testing will be performed within 2 weeks after hospital discharge.

The following main hypothesis will be tested:

- Combined assessment of coronary anatomy and myocardial perfusion using 320 MDCT results in a safe and optimized, cost-effective invasive treatment strategy

DETAILED DESCRIPTION:
MATERIAL

- Consecutive patients referred with chest pain in whom acute coronary syndrome has been excluded, yet with a maintained clinical suspicion of coronary artery disease will be included in the study. Only patients deemed clinically suited for subsequent invasive evaluation and treatment will be included.

METHODS

-If the patients accept participation in the trial a computerized 1:1 randomization for CTA alone (control group) or CTA and CTP combined (intervention group) within 2 weeks from discharge will be conducted. CT angiography and CT myocardial perfusion imaging will be performed using a 320-slice MSCT Toshiba VISION Edition Aquilion One scanner according to recommendations from the vendor and clinical routine developed at Rigshospitalet. Based on CTA and/or CTP findings patients will be referred for invasive evaluation including fractional flow reserve assessment (FFR) and treatment within 30 days. Invasive procedures will be performed according to international guidelines and the frequency of revascularization procedures recorded. Clinical outcome data according to specified secondary endpoints will be recorded from hospital charts and medical registries.

ELIGIBILITY:
Inclusion Criteria:

* Recent acute-onset chest pain where coronary artery disease is suspected
* During initial acute hospitalization:

  1. Normal coronary biomarkers (Troponins)
  2. No or non-diagnostic ECG changes (LV hypertrophy, bundle branch blok, pacemaker rhythm)
* Age ≥50 years
* ≥ 1 cardiovascular risk factor (family history of CAD, hypertension, hypercholesterolemia, diabetes, smoking) corresponding to a Duke clinical score ≥20%

Exclusion Criteria:

* Known Iodine contrast allergy
* Estimated GFR below 50 ml/min
* Adenosine intolerance - known allergic asthma
* Previous CABG
* Patient related circumstances which preclude informed consent from the patient
* Patients in whom psychiatric, physical or geographic conditions do not allow long-term clinical followup
* Expected survival of less that 2 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2013-10; Primary Completion 2017-03 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Frequency of coronary revascularization among included patients referred for invasive investigation | Within 60 days of study inclusion
  Among patients referred for invasive coronary evaluation the frequency of subsequent PCI and/or CABG is recorded

SECONDARY OUTCOMES:
Hospital admittance due to recurrence of chest pain, acute myocardial infarction or cardiac death | Within 3, 12 and 24 months after CT examination
New referral for invasive investigation following inititial evaluation | 3, 12 and 24 months after CT examination
Coronary revascularization - not including revascularization related to index evaluation | 3, 12 and 24 months after CT examination
Invasive procedure related events | Within 30 days of invasive procedure
  Among patients referred for invasive evaluation and treatment, procedure related events including death, bleeding, vascular complications, stroke and acute myocardial infarction will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Klaus F Kofoed, MD, DmSc, Principal Investigator — Department of Cardiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Denmark
Locations (7):
- Denmark (7):
  - Department of Cardiology and Radiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Copenhagen
  - Department of Cardiology, Amager University Hospital, Copenhagen
  - Department of Cardiology, Bispebjerg University Hospital, Copenhagen
  - Department of Cardiology, Gentofte University Hospital, Copenhagen
  - Department of Cardiology, Glostrup University Hospital, Copenhagen
  - Department of Cardiology, Herlev Hospital, Copenhagen
  - Department of Cardiology, Hvidovre University Hospital, Copenhagen

REFERENCES:
- [Background] Linde JJ, Kofoed KF, Sorgaard M, Kelbaek H, Jensen GB, Nielsen WB, Hove JD. Cardiac computed tomography guided treatment strategy in patients with recent acute-onset chest pain: results from the randomised, controlled trial: CArdiac cT in the treatment of acute CHest pain (CATCH). Int J Cardiol. 2013 Oct 15;168(6):5257-62. doi: 10.1016/j.ijcard.2013.08.020. Epub 2013 Aug 14. PMID 23998546
- [Background] Kuhl JT, Linde JJ, Fuchs A, Kristensen TS, Kelbaek H, George RT, Hove JD, Kofoed KF. Patterns of myocardial perfusion in humans evaluated with contrast-enhanced 320 multidetector computed tomography. Int J Cardiovasc Imaging. 2012 Oct;28(7):1739-47. doi: 10.1007/s10554-011-9986-z. Epub 2011 Dec 6. PMID 22143171